CLINICAL TRIAL: NCT01393119
Title: Phase II, Open-label, Loading and Maintenance Dose Finding Study of GTx-758 in Men With Prostate Cancer
Brief Title: Phase II, Dose Finding Study of GTx-758
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Clinical Hold
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G200710
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-fluoro-N-(4-fluorophenyl)-4-hydroxy-N-(4-hydroxyphenyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1000mg Loading Dose GTx-758 BID and Maintenance Dose 1000mg (Experimental): 1000mg Loading Dose GTx-758 BID and Maintenance Dose 1000mg
  Interventions: Drug: GTx-758
- 1000mg Loading DoseGTx-758 BID and Maintenance Dose 2000mg (Experimental): 1000mg Loading Dose GTx-758 BID and Maintenance Dose 2000mg
  Interventions: Drug: GTx-758
- 1500 mg Loading Dose GTx-758 BID and Maintenance Dose 1000mg (Experimental): 1500 mg Loading Dose GTx-758 BID and Maintenance Dose 1000mg
  Interventions: Drug: GTx-758
- 1500 mg Loading Dose GTx-758 BID and Maintenance Dose 2000mg (Experimental): 1500 mg Loading Dose GTx-758 BID and Maintenance Dose 2000mg
  Interventions: Drug: GTx-758

INTERVENTIONS:
Drug: GTx-758 — 3-fluoro-N-( 4-fluorophenyl)-4-hydroxy-N-( 4-hydroxyphenyl) benzamide; a nonsteroidal selective estrogen receptor (ER) a agonist

SUMMARY:
The purpose of this study is to determine the appropriate loading and maintenance dose of GTx-758 to reach and maintain castration for the duration of the study.

DETAILED DESCRIPTION:
The original purpose of the study was to determine the appropriate loading and maintenance dose of GTx-758 to reach and maintain castration for the duration of the study. The primary endpoint was used to assess the loading dose, while the secondary endpoint was intended to be used to assess maintenance. Due to the study being terminated early, as requested by FDA, the secondary assessment of maintenance was unable to be assessed. Hence, all summaries provided are for subjects in the two loading dose groups of 1000 mg BID and 1500mg BID only and not broken out by the maintenance dose.

ELIGIBILITY:
Inclusion Criteria:

1. Be between age 45 and 80 years of age
2. Be able to communicate effectively with the study personnel
3. ECOG is ≤2
4. Screening serum total testosterone ≥150 ng/dL
5. Have prostate cancer, confirmed by pathology report
6. Have not been treated with ADT (chemical or surgical). If a subject has been treated with LHRHa for ≤6 months duration and that treatment was ≥1 years prior to the screening, the subject may be considered for the study.
7. Have a clinical indication for the initiation ADT.
8. Give written informed consent prior to any study specific procedures
9. Subjects must agree to use acceptable methods of contraception:

   * If their female partners are pregnant or lactating acceptable methods of contraception from the time of the first administration of study medication until 3 months following administration of the last dose of study medication must be used. Acceptable methods are: Condom used with spermicidal foam/gel/film/cream/suppository. If the subject has undergone surgical sterilization (vasectomy with documentation of azospermia) a condom with spermicidal foam/gel/film/cream/suppository should be used.
   * If the male subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 3 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e. double barrier method of contraception], surgical sterilization (vasectomy with documentation of azospermia) and a double barrier method (condom used with spermicidal foam/gel/film/cream/suppository), the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a double barrier method (condom used with spermicidal foam/gel/film/cream/suppository).
   * If the female partner has undergone documented tubal ligation (female sterilization), a double barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used.
   * If the female partner has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a double barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used.

Exclusion Criteria:

1. Known hypersensitivity or allergy to estrogen or estrogen like drugs
2. Have, in the judgment of the Investigator, a clinically significant concurrent illness or psychological, familial, sociological, geographical or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol
3. History of abnormal blood clotting, Factor V Leiden clotting disorder, thrombotic disease (venous or arterial thrombotic events such as history of myocardial infarct (MI), stroke, deep vein thrombosis (DVT), and/or pulmonary embolus (PE)) NOTE: if there is evidence of an MI on the ECG that is not documented in the medical history or there is a history of MI greater than three years ago that has completely resolved, the eligibility of this subject per this exclusion criterion is an investigator decision and may require a consultation with a cardiologist.
4. Have ALT or AST above 2 times the upper limit of normal (ULN)
5. Have alkaline phosphatase greater than 3 times ULN and/or total bilirubin levels above 2 mg/dL at baseline
6. Patients cannot have brain or spinal cord metastases
7. Patients cannot have or be at high risk for spinal cord compression from bone metastases.
8. Received an investigational drug within a period of 90 days prior to enrollment in the study
9. Received the study medication previously
10. Currently taking testosterone, testosterone-like agents or antiandrogens, including 5-alpha reductase inhibitors (the subject may be considered for randomization after a 4 week washout period prior to randomization)
11. Currently taking Saw Palmetto or PC-SPES (the subject may be considered for randomization after a 4 week washout period prior to randomization)
12. Have taken diethylstilbestrol or other estrogen products within the previous 12 months prior to randomization into this study
13. Have taken body building or fertility supplements within 4 weeks of admission into the study (steroids and steroid like supplements)
14. Have a history of cancer other than prostate cancer, superficial bladder cancer (with no recurrence in the last 5 years) and/or non-melanoma carcinoma of the skin.
15. QTcB >480 msec, If the first QTcB reading exceeds 480 msec two additional ECGs are to be performed separated at least 5 min apart, then take the average of the three QTcB readings to determine if the subject satisfies the above criteria. If the average QTcB reading is > 480 msec then the subject is excluded.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Steiner, MD, Study Director — GTx
Locations (21):
- United States (21):
  - GTx Investigative Site, Glendale, Arizona
  - GTx Investigative Site, Phoenix, Arizona
  - GTx Investigative Site, La Mesa, California
  - GTx Investigative Site, San Bernardino, California
  - GTx Investigative Site, Aventura, Florida
  - GTx Investigative Site, Bradenton, Florida
  - GTx Investigative Site, St. Petersburg, Florida
  - GTx Investigative Site, Tampa, Florida
  - GTx Investigative Site, Roswell, Georgia
  - GTx Investigative Site, Jeffersonville, Indiana
  - GTx Investigative Site, Shreveport, Louisiana
  - GTx Investigative Site, Annapolis, Maryland
  - GTx Investigative Site, Towson, Maryland
  - GTx Investigative Site, Hamilton, New Jersey
  - GTx Investigative Site, Albany, New York
  - GTx Investigative Site, Oneida, New York
  - GTx Investigative Site, Syracuse, New York
  - GTx Investigative Site, Concord, North Carolina
  - GTx Investigative Site, Cincinnati, Ohio
  - GTx Investigative Site, Columbus, Ohio
  - GTx Investigative Site, Bala-Cynwyd, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 patients were screened with 19 discontinuing the study due to screen failure. 77-19=58 randomized subjects. Please note, 3 of these 58 subjects were randomized but not treated, as noted below, hence n=55 subjects are provided data for results summaries.
  Note: Due to study being terminated early, per FDA, secondary assessment of maintenance was not assessed. Hence, all summaries are for the two loading dose groups of 1000 mg BID and 1500mg BID only.
Pre-assignment Details: Screen Failure subjects were not included in the outputs from the previous company who owned the product.
Groups:
- Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758: Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758
- Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758; Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758: Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758
- Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758: Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758
Period: Overall Study
Arm/Group | Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758 | Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758 | Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758 | Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758
Started | 14 | 14 | 14 | 16
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 14 | 14 | 16
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Randomized but Not treated | 1 | 0 | 1 | 1
Not completed — Sponsor Termination of Study | 11 | 12 | 9 | 12

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758: Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758
- Total: Total of all reporting groups
Arm/Group | Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758 | Loading Dose 1000mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758 | Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 1000mg GTx-758 | Loading Dose 1500mg GTx-758 BID and Maintenance Dose of 2000mg GTx-758 | Total
Number analyzed (Participants) | 13 | 14 | 13 | 15 | 55
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age, Continuous | 64.8 (4.9) | 67.1 (8.4) | 68.0 (5.4) | 68.9 (8.2) | 67.25 (6.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males | 13 | 14 | 13 | 15 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 14 | 13 | 13 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 5 | 13
  White | 11 | 10 | 9 | 10 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That Reach Castration by Day 28
Description: Percentage of Patients Note: Due to the study being terminated early, per FDA, the secondary assessment of maintenance was unable to be assessed. Hence, all summaries provided are for subjects in the two loading dose groups of 1000 mg BID and 1500mg BID only.
  PLEASE NOTE: Study was terminated early, per FDA, the secondary assessment of maintenance was unable to be assessed. Hence, the efficacy summary provided are for subjects in the two loading dose groups of 1000 mg BID and 1500mg BID only, poling across maintenance doses within each loading dose.
  Safety/ITT - 27 and 28 patients, respectively mITT - 18 and 19 patients, respectively Note: mITT includes patients that meet the requirements for the efficacy analyses
  This format was agreed to by the PRS review team, per email communication on guidnace for presenting the data.
Time Frame: Day 1-28
Population: Modified Intent to Treat Population
Measure: Count of Participants; unit: Participants
Groups:
- 1000mg GTx-758 BID: Loading dose 1000mg GTx-758 BID + maintenance dose of 1000mg/2000mg GTx-758 daily Combined
- 1500 mg GTx-758 BID: Loading dose of 1500 mg GTx-758 BID + maintenance dose of 1000mg/2000mg GTx-758 daily Combined
Arm/Group | 1000mg GTx-758 BID | 1500 mg GTx-758 BID
Number analyzed (Participants) | 18 | 19
Participants | 15 | 16

ADVERSE EVENTS:
Groups:
- 1000mg GTx-758 BID: Loading dose 1000mg GTx-758 BID + maintenance dose of 1000mg GTx-758 daily
- 1000 mg GTx-758 BID: Loading dose of 1000mg GTx-758 BID + maintenance dose of 2000mg GTx-758 daily
- 1500 mg GTx-758 BID: Loading dose of 1500 mg GTx-758 BID + maintenance dose of 1000mg GTx-758 daily
- 1500mg GTx-758 BID: Loading dose of 1500mg of GTx-758 BID + maintenance dose of 2000mg GTx-758 daily
Arm/Group | 1000mg GTx-758 BID | 1000 mg GTx-758 BID | 1500 mg GTx-758 BID | 1500mg GTx-758 BID
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/13 | 1/15
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/14 | 0/13 | 3/15
Other Adverse Events (participants affected / at risk) | 10/13 | 12/14 | 10/13 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1000mg GTx-758 BID (N=13) | 1000 mg GTx-758 BID (N=14) | 1500 mg GTx-758 BID (N=13) | 1500mg GTx-758 BID (N=15)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
DVT (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1000mg GTx-758 BID (N=13) | 1000 mg GTx-758 BID (N=14) | 1500 mg GTx-758 BID (N=13) | 1500mg GTx-758 BID (N=15)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 3
Fatigue (General disorders) | 4 | 1 | 1 | 4
Influenza Like Illness (General disorders) | 2 | 0 | 1 | 0
Odema Peripheral (General disorders) | 0 | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 2 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Breast Pain (Reproductive system and breast disorders) | 5 | 1 | 2 | 3
Gynaecomastia (Reproductive system and breast disorders) | 0 | 2 | 2 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
DVT (Vascular disorders) | 2 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 1 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No